CLINICAL TRIAL: NCT00296946
Title: Phase II Clinical Trial of Ipratropium Bromide Spray as a Treatment for Sialorrhea in Patients With Parkinson's Disease
Brief Title: Ipratropium Spray for Drooling Saliva in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Parkinson's Disease Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FY2005
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2004-10

CONDITIONS: Parkinson's Disease
Keywords: Sialorrhoea
MeSH Terms: conditions — Parkinson Disease; Sialorrhea | interventions — Ipratropium; Pharmaceutical Preparations

INTERVENTIONS:
Drug: ipratropium bromide (drug)

SUMMARY:
A phase II double blind clinical trial investigating the effects of ipratropium spray versus placebo spray in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Background: Excessive drooling of saliva (sialorrhoea) is a common complication of Parkinson's disease (PD). Unfortunately current medications, which rely on anticholinergic properties, often induce systemic side effects, such as confusion, hallucinations or urinary retention.

Aim: We therefore hypothesise that local application of an anticholinergic aerosol spray into the mouth would reduce sialorrhea in PD without inducing systemic side-effects.

Method: A double blind, randomised, placebo-controlled cross-over trial of the muscarinic antagonist, ipratropium bromide in patients with bothersome drooling in idiopathic Parkinson's disease. All patients are recruited from the Movement Disorders Clinic, Toronto Western Hospital and informed consent is obtained. Patients are randomised to receive ipratropium bromide, 1- 2 metered doses (sprays) of active drug (21 micorgram per metered dose) or matching placebo, up to a maximum of 4 times per day, in a double-blind, cross-over design using randomisation tables. Total treatment length is two weeks for each limb of the study with a 1-2 week wash out period. The primary outcome measure is an objective measure of saliva production. Dental rolls are inserted into the mouth for 5 min and the patient instructed not to swallow and sit upright. The weight of dental rolls before and after insertion is calculated as a measure of saliva production. The secondary outcome measures are subjective measure of saliva where patients or caregivers record the level of saliva production each day for the 2 weeks of each treatment using validated subjective rating scales which assess drooling severity and frequency. In addition, parkinsonism is rated using the UPDRS parts I - IV and adverse events are recorded. The scores for measured saliva production following ipratropium bromide and placebo treatment will be compared using appropriate paired t-tests. Results from the scales assessing the subjective measures of saliva production and UPDRS ratings will be compared via paired non-parametric Wilcoxon matched pairs test. 20 patients will be recruited.

ELIGIBILITY:
Inclusion Criteria:Male and female patients with idiopathic PD and who are currently experiencing bothersome drooling (United Parkinson's Disease Rating Scale (UPDRS) item 6, rating of 2 or higher) will be eligible for this study. Patients must be on a stable medication regimen for the preceding one-month run-in period. In addition, patients or a caregiver must be able to complete a daily record card, and patients must be able to tolerate an oral dental roll for 5-minute periods for saliva measurements.

-

Exclusion Criteria:

Patients taking acetylcholinesterase inhibitors, cholinergic agents, or anticholinergic agents, history of glaucoma, clinically significant urinary outflow obstruction or urinary retention, active psychosis or hallucinations, and allergy to peanuts or soybeans. -

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2004-11; Study Completion 2006-06

PRIMARY OUTCOMES:
objective measure of saliva production.

SECONDARY OUTCOMES:
subjective measure of saliva using diaries
UPDRS parts I - IV
adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Fox, MRCP, PhD, Principal Investigator — University Health Network, Toronto, Canada
Locations (1):
- Toronto Western Hospital, University Health Network, Toronto, Ontario, Canada